CLINICAL TRIAL: NCT06091280
Title: Home-Based Respiratory Muscle Strength Training Program for Individuals With Post-COVID-19 Persistent Dyspnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 006272
Record Dates: First submitted 2023-10-18; First posted 2023-10-19 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Post-COVID-19 Syndrome; Dyspnea
Keywords: Respiratory muscle strength training; Respiratory symptoms
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Dyspnea; Signs and Symptoms, Respiratory

STUDY DESIGN:
Intervention Model Description: Single-group, longitudinal, intervention study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Respiratory Muscle Strength Training (Experimental): Pursed Lip Breathing: Participants will perform two sets of 10 repetitions twice per day.
  Inspiratory Muscle Strength Training (IMST): The participant will use an IMST trainer provided by the study (Threshold Inspiratory Muscle Strength Trainer). This exercise is repeated for a 3-minute duration, followed by a rest period of 2 minutes. This cycle is repeated for 6 cycles over a 30-minute timespan. This exercise will be performed 3 times/week on alternating days.
  Expiratory Muscle Strength Training (EMST): The participant will use an EMST trainer (EMST 150) provided by the study. This exercise is repeated for a 3-minute duration, followed by a rest period of 2 minutes. The cycle is repeated for 6 cycles over a 30-minute timespan. This exercise will be performed 3 x/week on opposite days of the inspiratory muscle strength training.
  Interventions: Device: Respiratory Muscle Strength Trainers

INTERVENTIONS:
Device: Respiratory Muscle Strength Trainers — Devices provided to each participant. Resistance loading set at less than 50% of the peak inspiratory and peak expiratory flow rate.
  Other Names: Threshold Inspiratory Muscle Strength Trainer; Expiratory Muscle Strength Trainer (EMST 150)

SUMMARY:
To evaluate the extent to which a 12-week respiratory rehabilitation program consisting of inspiratory and expiratory breathing exercises compared to expiratory breathing exercises alone will help to improve shortness of breath, respiratory symptoms, breathing function, distance walked, and quality of life in those who are experiencing persistent shortness of breath after having had COVID-19. Measurements will take place at the beginning, 6 weeks, and at 12 weeks in the study.

DETAILED DESCRIPTION:
To evaluate the extent to which a 12-week respiratory rehabilitation program consisting of inspiratory and expiratory muscle strength training exercises as compared to a prior study of expiratory muscle strength training alone is effective in improving dyspnea, respiratory symptoms, quantitative measures of pulmonary function, physical performance, and quality of life in individuals reporting persistent dyspnea post-COVID-19 at baseline, six and twelve weeks.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported history of a positive COVID-19 diagnosis in the past.
* Able to walk independently
* Cognitively intact
* English-speaking
* Dyspnea at rest or with activity rated at 3 or greater on the Dyspnea on Exertion scale.
* May use oxygen.
* May be taking medications.

Exclusion Criteria:

* Individuals who are wheelchair bound or who cannot walk independently.
* Individuals hospitalized for COVID-19 who self-report that they received mechanical ventilation during hospitalization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-12-23 (Actual); Study Completion 2025-03-14 (Actual)

PRIMARY OUTCOMES:
Modified Medical Research Council Scale | Baseline, 6-weeks, and 12-week measurements
  Scale of 0-4 with 4 being the most severe dyspnea.
COPD Assessment Test | Baseline, 6-weeks, and 12-week measurements.
  8-item questionnaire with a semantic, 6-point differential scale for each item. Scores range from 0-40 with higher scores indicating more severe respiratory symptoms.
Forced Expiratory Volume over 1 second (FEV1) | Baseline, 6-weeks, and 12-week measurements
  Using the Microlife Digital Peak Flow and FEV1 Meter (Clearwater, FL).
Peak Inspiratory Flow | Baseline, 6-weeks, and 12-week measurements.
  Using the In-Check Peak Inspiratory Flow meter (Granbury, TX).
Thoracic Expansion Measures | Baseline, 6-weeks, and 12-week measurements
  Gulick tape measure positioned around the participant's chest at the 4th intercostal space. Participant breathes in and out as far as possible and the difference between the 2 values equals thoracic expansion.
Physical Capacity | Baseline, 6-weeks, and 12-week measurements.
  6 Minute Walk Test following the American Thoracic Society Procedure: 50-meter distance is marked. Participant walks as quickly as possible for 6 minutes. Results recorded in meters. Vital signs and oxygen saturation monitored and recorded.
EuroQoL-5 Dimension-5 Level | Baseline, 6-weeks, and 12-week measurements.
  EuroQoL-5 Dimension-5 Level to evaluate 5 dimensions of quality of life including mobility, self-care, usual activities, discomfort and pain, anxiety, and depression. Each is scored using a 5-point semantic scale.

SECONDARY OUTCOMES:
Feasibility and Acceptability of the Intervention | 12-weeks.
  Recruitment and retention rates. 5-item questionnaire asking participants about the exercise protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Constance Visovsky, PhD, Principal Investigator — University of South Florida
Locations (1):
- University of South Florida, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be available at the end of the study to other investigators and will include the data associated with the study outcomes (Dyspnea, quality of life, pulmonary symptoms, thoracic expansion, pulmonary function tests, six minute walk test, demographics, and feasibility and acceptability).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available following publication of the study outcomes, and for a period of one year.
Access Criteria: A formal request to the primary investigator (Dr. Constance Visovsky).

REFERENCES:
- [Background] Borg GA. Psychophysical bases of perceived exertion. Med Sci Sports Exerc. 1982;14(5):377-81. PMID 7154893
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Jones PW, Harding G, Berry P, Wiklund I, Chen WH, Kline Leidy N. Development and first validation of the COPD Assessment Test. Eur Respir J. 2009 Sep;34(3):648-54. doi: 10.1183/09031936.00102509. PMID 19720809
- [Background] Mahler DA, Wells CK. Evaluation of clinical methods for rating dyspnea. Chest. 1988 Mar;93(3):580-6. doi: 10.1378/chest.93.3.580. PMID 3342669
- [Background] Morgan S, Visovsky C, Thomas B, Klein AB, Ji M, Schwab L, Coury J. Home-Based Pilot Pulmonary Program for Dyspneic Patients Post-COVID-19. Clin Nurs Res. 2023 Jun;32(5):895-901. doi: 10.1177/10547738231170496. Epub 2023 May 3. PMID 37132243
- [Background] Mota S, Guell R, Barreiro E, Solanes I, Ramirez-Sarmiento A, Orozco-Levi M, Casan P, Gea J, Sanchis J. Clinical outcomes of expiratory muscle training in severe COPD patients. Respir Med. 2007 Mar;101(3):516-24. doi: 10.1016/j.rmed.2006.06.024. Epub 2006 Aug 30. PMID 16942867
- [Derived] Morgan SP, Thomas B, Rodriguez CS, Johnson A, Beckie TM. Inspiratory and Expiratory Muscle Strength Training for Persistent Dyspnea in Post-COVID-19. Clin Nurs Res. 2025 Nov;34(8):462-471. doi: 10.1177/10547738251371244. Epub 2025 Sep 25. PMID 40995943